CLINICAL TRIAL: NCT04969965
Title: A Single Dose Phase 1 Study in Healthy Participants to Evaluate the Comparative Pharmacokinetics of Orally Administered EQ143 in Different Racial and Ethnic Populations
Brief Title: To Evaluate the Comparative Pharmacokinetics of Orally Administered EQ143 in Different Racial and Ethnic Populations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EQRx, Inc. (Industry)
Responsible Party: Sponsor
Organization: EQRx International, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQ143-101
Record Dates: First submitted 2021-07-13; First posted 2021-07-21 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: NSCLC; Healthy Volunteers; Pharmacokinetics
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aumolertinib (Experimental): single dose oral 110mg of aumolertinib
  Interventions: Drug: aumolertinib

INTERVENTIONS:
Drug: aumolertinib — EQ143 tablet is an oral solid dosage form manufactured at a strength of 55 mg
  Other Names: EQ143

SUMMARY:
This is an open-label and uncontrolled study to evaluate the comparative PK of EQ143 following oral single dose administration in adult healthy volunteers different racial and ethnic populations.

A total of one (1) single dose cohort is planned at 110 mg of EQ143. EQ143 is an approved therapy in China at the 110 mg dose for the treatment of patients with Epidermal Growth Factor Receptor (EGFR) T790Mmutation-positive, metastatic non-small cell lung cancer (NSCLC), who have progressed during or after EGFR tyrosine kinase inhibitor (TKI) therapy.

A total of 45 (15 Caucasian, 8 Black/African American and 7 Hispanic/Latino, and 15 ethnic Chinese)

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a participant has to meet all of the following inclusion criteria:

1. Participant self-reports as being of one of the following racial or ethnic groups:

   1. being of non-Chinese, European descent
   2. having origins in any of the black racial groups of Africa
   3. being of Cuban, Mexican, Puerto Rican, Cuban, South or Central American, or other Spanish culture or origin, regardless of race
   4. having two Han Chinese biological parents;
2. Is capable of giving informed consent and complying with study procedures;
3. Healthy male or female participants, between the ages of 18 and 65 years, inclusive at the time of informed consent;
4. Body mass index (BMI) of 18.0 to 34.9 kg/m2 inclusive and body weight not less than 50 kg;
5. Female participants must have a negative serum pregnancy test result at Screening and negative urine pregnancy test at admission to the study site, are not currently breastfeeding, and meet one of the following criteria:

   1. Surgically sterile for at least 3 months prior to Screening by one of the following means:

      * Bilateral tubal ligation
      * Bilateral salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   2. Postmenopausal, defined as the following:

      * Last menstrual period greater than 12 months prior to Screening without an alternative medical cause, AND
      * Postmenopausal status confirmed by serum Follicle-stimulating hormone (FSH) concentration at Screening > 40 mIU/mL
   3. Female participants of childbearing potential must use at least one of the following protocol-specified highly effective methods of birth control, AND must agree to use barrier contraception (male condom) during heterosexual intercourse, from the time of Screening until at least 90 days after EQ143 treatment:

      * Infertile male partner (eg, vasectomy [at least 6 months prior to Screening; vasectomized partner should be the sole partner of the female participant], permanently sterile following bilateral orchidectomy, or any other documented cause of infertility)
      * Combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal, injectable)
      * Progestogen-only hormonal contraception (oral, injectable, implantable)
      * Implantable device (implantable rod or intrauterine device)
      * Bilateral tubal occlusion Alternatively, females of childbearing potential must practice complete abstinence (defined as refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the participant; periodic abstinence and withdrawal are not acceptable) from Screening until at least 90 days after EQ143 treatment. It is not necessary to use any other method of contraception when complete abstinence is elected. Women of childbearing potential (WOCBP) who choose complete abstinence must continue to have pregnancy tests as per protocol. The reliability of sexual abstinence needs to be evaluated by the Investigator in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

   Participants must agree to not donate sperm or ova from time of EQ143 administration until 90 days after EQ143 treatment.
6. Male participants must agree to utilize a highly effective method of contraception (condom) during heterosexual intercourse from CRU admission until 12 weeks following the final Follow-up visit on Day 10 and must refrain from donating sperm for this same period;
7. Considered healthy by the Investigator, based on participant's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center;
9. Participants willing to defer receiving prophylactic live immunizations during the duration of the study. Participants may receive vaccination for SARS-CoV-2 at the discretion of the Investigator as soon as they are eligible, and a vaccine is available. If and when possible, the inactivated mRNA-based vaccines are recommended.

Exclusion Criteria:

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. Inability to attend all the study visits or comply with study procedures;
2. Evidence of clinically significant history of gastrointestinal, musculoskeletal, endocrine, hematologic, renal, hepatic, neurologic, ophthalmic, immunologic, lipid metabolism disorders, drug hypersensitivity, psychiatric disease and abnormalities or any known history of any gastrointestinal surgery or cholecystectomy that could impact the PK of EQ143 as determined by the Investigator or Sponsor;
3. Evidence of clinically significant history of cardiovascular disease, including myocardial infarction, unstable angina, Torsade de Pointes, clinically significant arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), symptomatic congestive heart failure (New York Heart Association class III or IV), cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism or other clinically significant episode of thromboembolic disease;
4. A history of additional risk factors for Torsade de Pointes (eg, heart failure, hypokalemia, family history of Long QT Syndrome);
5. Evidence of clinically significant history of bronchopulmonary disease, including interstitial lung disease (ILD), drug induced ILD, radiation pneumonia requiring steroid treatment and clinical evidence of active ILD;
6. Female participants of childbearing potential except as permitted by 5 a, b, or c under inclusion criteria;
7. Hospital admission or major surgery within 3 months prior to Screening;
8. A history of prescription drug abuse, or illicit drug use within 6 months prior to Screening;
9. A history of alcohol abuse according to medical history within 6 months prior to Screening;
10. A history of organ transplant, including history of bone marrow transplant;
11. Taken any prescription medications (excluding contraceptives) within 14 days or 5 half-lives (whichever is longer) of the study dose or taken an investigational drug within 3 months or 5 half-lives, whichever is longer, from the Screening date;
12. Evidence of hypertension stage 2, defined as a systolic BP > 140 mmHg and a diastolic BP > 90 mmHg at Screening. Blood pressure measurement should be performed in triplicate if initial results exceed these values, and the average value should be used to determine eligibility;
13. Fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening. PCR testing for SARS-CoV-2 infection will be performed in accordance with local guidelines (health authorities, Institutional Review Boards/Independent Ethics Committees, and study center policies) and at the discretion of the Investigator, if required;
14. Any of the following ECG criteria at Screening or Admission:

    1. PR interval > 220 ms or < 110 ms;
    2. QRS interval > 120 ms;
    3. QTcF interval > 450 ms in males and > 480 ms in females;
    4. A marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval > 450 ms)
    5. ST segment elevation or depression considered to be clinically significant by the Investigator or designee;
    6. T-wave abnormalities considered to be clinically significant by the Investigator or designee; If the QTcF interval exceeds 450 ms (males) or 480 ms (females), or the QRS interval exceeds 120 ms, the ECG should be repeated in triplicate and the average of the 3 QTcF or QRS values should be used to determine the patient's eligibility.
15. Impaired renal function as determined by Investigator following review of clinical laboratory test results (ie, estimated glomerular filtration rate [eGFR] less than 90 mL/min/1.73m2, as calculated using the method standard for the institution);
16. Any of the following safety laboratory findings at Screening or Admission:

    1. Absolute neutrophil count < 1.5 × 109/L
    2. Platelet count < 100 × 109/L
    3. Hemoglobin < 90 g/L (< 9 g/dL)
    4. International Normalized Ratio (INR) > 1.5
    5. Creatinine outside normal limits
17. Positive blood screen for HIV, positive Hepatitis B core antibody (HBcAb) and positive Hepatitis B surface antigen (HBsAg), positive Hepatitis C virus antibody (HCV Ab) and positive HCV polymerase chain reaction (PCR), positive Hepatitis A antibody. Note: A positive HCV Ab with negative HCV PCR, positive HBcAb with negative HBsAg, positive Hepatitis A virus with negative immunoglobulin M (IgM) will be eligible;
18. Participants with major clinical infections within 3 months prior to Screening or any symptoms of infection within 7 days prior to Screening (not applicable to participants with cutaneous fungal infection);
19. Participants who have received live vaccines or attenuated vaccines within 1 month before dosing. Participants may receive vaccination for SARS-CoV-2 at the discretion of the Investigator as soon as they are eligible and a vaccine available. If and when possible, the inactivated mRNA-based vaccines are recommended;
20. Donated or lost > 500ml of blood in the previous 3 months prior to Screening;
21. Any liver function panel analyte (LFT) value > 1.5 × upper limits of normal reference range (ULN) which includes aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline Phosphatase (ALP), and gamma-glutamyl transferase (GGT) at Screening or at Admission. Bilirubin should be > ULN, or > 3 × ULN for participants with well-documented Gilbert's Syndrome;
22. Participants who have taken a special diet (including dragon fruit, mango, grapefruit, starfruit, Seville oranges etc.) or other factors affecting drug absorption, distribution, metabolism, and excretion within 48 hours before taking EQ143;
23. Use of prescription medications (excluding contraceptives) within 14 days, over the counter (OTC) medication within 7 days, and herbal supplements, dietary supplements, protein powders, and fish oil within 7 days prior to dosing (Note: Use of acetaminophen/paracetamol at < 2 g/day is permitted until 24 hours prior to dosing. Any other nonsteroidal anti-inflammatory drugs [NSAIDs]/antihistamines if permitted can be discussed on a case-by-case basis by the Medical Monitor [MM] and Sponsor). Prophylactic medication may continue as long as this is approved by the MM and Sponsor prior to inclusion;
24. Participants who have dysphagia or any history of gastrointestinal diseases that affect drug absorption or have undergone operations that affect drug absorption;
25. Participants with any other active malignancy within 5 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ;
26. Any condition or finding that in the opinion of the Principal Investigator or designee would put the participant or study conduct at risk if the participant were to participate in the study.
27. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the Follow-up period.
28. Participants who are regular smokers, ie, smoke more than five cigarettes per day or more than 10 packets per year and are not willing to refrain from smoking from 48 hours before EQ143 administration through to the final Follow-up visit on Day 10.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
To compare the concentration (called PK) of EQ143 in the blood following a single oral administration in adult, healthy participants. | Pharmacokinetic (PK) blood sampling will be conducted at pre-dose (within 1 hour prior to dosing) on day 1at an interval of 1 and 2 hours and Day 2, Day 3, Day 4, Day 5, Day 6, and Day 8 post-dose and at the end of study (EOS) visit (10 days post-dose).

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of EQ143 following a single oral administration in adult, healthy, Caucasian, Black or African American, Hispanic or Latino, and ethnic Chinese populations. | 12-38 Days

CONTACTS AND LOCATIONS:
Locations (2):
- Spaulding Clinical Research, West Bend, Wisconsin, United States
- New Zealand Clinical Research, Auckland, New Zealand